CLINICAL TRIAL: NCT06042127
Title: Per-oral Endoscopic Myotomy With Fundoplication for Achalasia - an International Multicenter Randomized Controlled Trial
Brief Title: POEM-F for Achalasia International Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Deenanath Mangeshkar Hospital and Research Centre (Other); Johns Hopkins University (Other); Northwestern University Feinberg School of Medicine (Other); Nanfang Hospital, Southern Medical University (Other); Asian Institute of Gastroenterology, India (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023 145-T
Record Dates: First submitted 2023-09-06; First posted 2023-09-18 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Achalasia
Keywords: POEM; Fundoplication; GERD
MeSH Terms: conditions — Esophageal Achalasia; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Per-oral endoscopic myotomy with fundoplication (Experimental): The detail of the procedure has been reported in the literature. After completion of myotomy as per conventional anterior POEM, a serosal incision would be made at the level of the GE junction below the diaphragmatic crus. The peritoneal cavity would then be entered and the anterior gastric wall could be identified. A detachable endoloop would be introduced alongside the endoscope with the guidance of endoscopic clip. Three to four clips would be applied to the anterior gastric fundus while additional 3-4 clips would be applied to the edge of the submucosal tunnel, all anchoring to the endoloop. Upon tightening of the endoloop the anterior fundus would be approximated to the esophagogastric junction and thus completing the partial anterior fundoplication. Abdominal paracentesis to treat capnoperitoneum would be performed as required based on patient's clinical condition.
  Interventions: Procedure: POEM-F
- Conventional POEM (Active Comparator): Conventional per-oral endoscopic myotomy An anterior POEM would be performed per usual manner described in the literature. The procedure would be performed under general anaesthesia by expert endoscopists with at least 50 case experience of conventional POEM and 5 cases experience of POEM-F. The requirement of POEM experience is based on a recent multicenter study of learning curve by Fujiyoshi Y, et al. The procedure would follow the current recommendations from expert panel in reducing GER, including avoidance of excessive gastric myotomy and preservation of the sling fibers are the gastric cardia. The length of the esophageal and gastric myotomy is standardized at 5cm and 2cm respectively
  Interventions: Procedure: Conventional POEM

INTERVENTIONS:
Procedure: POEM-F — POEM-F would be performed as described in the arms section
  Arms: Per-oral endoscopic myotomy with fundoplication
Procedure: Conventional POEM — Anterior POEM performed as described in the arms section
  Arms: Conventional POEM

SUMMARY:
Per-oral endoscopic myotomy (POEM) has emerged as the endoscopic treatment of choice for achalasia, offering comparable symptom relief with laparoscopic Heller's cardiomyotomy. The main concern with POEM is the higher incidence of post-procedure gastroesophageal reflux disease (GERD), occurring in up to 50-60% of patients. In order to reduce the risk of GERD, endoscopic fundoplication has been developed as a novel procedure mimicking surgical anterior partial fundoplication that can be performed in the same session as POEM (POEM-F). Case series of POEM-F in patients with achalasia reported encouraging outcomes of low GERD rate of ~12% at 1 year. Prospective comparative data between POEM-F and conventional POEM on post-procedure GERD is current lacking. The investigators therefore designed an international multicenter prospective randomized study to investigate the efficacy of POEM-F. The investigators postulate that POEM-F could reduce the incidence of post-procedure GERD when compared with conventional POEM.

This is an international multicenter randomized controlled trial conducted between high volume expert centers from Hong Kong SAR, China, India and United States of America. Adult patients with manometry confirmed achalasia would be randomised to undergo POEM-F or POEM. The procedure would be performed by experts with vast experience in POEM. The primary outcome is the incidence of post-procedure GERD at 1 year, defined by the updated Lyon consensus. Secondary outcomes include technical and clinical success rates, adverse events, post-POEM endoscopic and manometry findings as well as patients' symptom scores.

Sample size calculation Based on existing pilot comparative data on POEM-F and POEM, it is estimated that 84 patients would be required to demonstrate a difference in post-procedure GERD of 47.6% to 18.2%, with 80% power and false positive rate of 0.05, accounting for 10% loss to follow-up.

Purpose and potential The current study proposal could demonstrate the superiority of POEM-F over POEM in reducing post-procedural GERD. It would also demonstrate the safety and reproducibility of the technique in expert centers across the globe. It could potentially replace conventional POEM as the preferred minimally invasive endoscopic treatment for achalasia.

DETAILED DESCRIPTION:
Achalasia is the most common esophageal motility disorder worldwide, with an annual incidence of 1.6 per 100'000 individual and prevalence of 10 per 100'000 population. The incidence of achalasia has been dramatically rising over the past decade. A study conducted in Chicago suggested that over the 10 years from 2004 to 2014, the incidence and prevalence of achalasia were two- to threefold greater than estimates would have predicted. The likely explanation to the rise in incidence is an increased awareness of this condition and widespread availability of accurate diagnostic test with high resolution manometry. The cardinal features of achalasia include failed relaxation of lower esophageal sphincter and absent esophageal peristalsis. Owing to the benign nature of the disease, patients suffering from it would experience longstanding debilitating symptoms of dysphagia, chest pain, regurgitation, resulting in poor quality of life. In the past, laparoscopic Heller's cardiomyotomy with partial fundoplication and endoscopic pneumatic dilatation were considered as treatment options for achalasia.

In the past 10 years, per-oral endoscopic myotomy (POEM) has emerged as the incisionless minimally invasive endoscopic treatment of choice for achalasia. This Natural Orifice Transluminal Endoscopic Surgical (NOTES) technique involves mucosal incision and creation of a submucosal tunnel in the distal esophagus down to gastric cardia, followed by esophageal and gastric myotomy. Since the procedure was first reported by Inoue H, et al in 2010, it has seen worldwide acceptance as first-line therapy. POEM has been associated with excellent relief of dysphagia and achalasia-related symptoms with a low and acceptable adverse event rate of 0.5%. In a previous randomised controlled trial, POEM had a higher treatment success rate than pneumatic dilatation. When compared with laparoscopic Heller's cardiomyotomy, POEM was associated with at least similar treatment efficacy and a trend towards reduced short term adverse event. POEM could perform even better than surgical myotomy in patients with type III achalasia.

The main limitation of POEM is the incidence of gastroesophageal reflux disease (GERD) post-POEM. Kumbhari et al. looked at rates of GERD after POEM on patients who underwent subsequent objective pH testing. A total of 282 patients were included in this analysis from multiple centers in America, Asia, and Europe. About 58% of patients had objective evidence of abnormal acid exposure, with 23% showing evidence of esophagitis. More concerning, however, was that 60% of the patients with GERD were completely asymptomatic. This highlights an important issue at hand that many patients, either related to the propensity of GERD to be silent or the nature of achalasia to develop and insensate esophagus, do not report symptoms while showing high rates of GERD. POEM has been found to be consistently associated with higher rate of GERD than conventional Heller's cardiomyotomy or pneumatic dilatation across multiple studies.

Supported by evidence demonstrating the efficacy of partial fundoplication during Heller's operation, there has been a significant interest in performing fundoplication after POEM during the same session to prevent the development of post-POEM GERD. Inoue et al. pioneered the technique of POEM-F that mimics the surgical Dor (anterior partial fundoplication) procedure. In the pilot study, technical success was achieved in all 21 patients, and all but one had an intact fundoplication wrap on upper endoscopy at a 1-month follow-up. Four more studies conducted in Japan and India have reported good early outcomes with POEM-F (Technical success of 85-100%) for achalasia. No severe adverse event has been reported in these studies which reiterates the safety of this procedure. In the longest follow-up study on POEM-F, GERD diagnosed by an abnormal esophageal acid exposure was seen in 11.1% of the 21 cases at one-year follow-up: comparable (8.8%) to a large meta-analysis of 4871 Heller's cardiomyotomy with fundoplication procedures.

To date, no prospective multicenter randomised study has been conducted to compare the efficacy of POEM-F with conventional POEM in reducing post-procedure GERD. Therefore, in this study, the investigators aim to evaluate the of POEM-F in patients with achalasia through an international multicenter randomized controlled trial.

ELIGIBILITY:
Inclusion criteria:

1. Adult patient (age ≥18 and ≤65 years-old) and with symptomatic achalasia type I or II.
2. Capability of understanding and complying with the study requirements, including filling the Eckardt Score, GERD-HRQL and RSI questionnaire and signing the informed consent form.
3. Patients with achalasia type I, II or III who are one of the following:

   * Treatment naïve, or
   * Failed prior through-the-scope balloon dilation, Savary or pneumatic dilation

Exclusion criteria:

1. Patients unable or unwilling to provide consent.
2. Previous esophageal or gastric surgery.
3. Prior achalasia treatment including Heller myotomy, POEM.
4. Sigmoid achalasia, or significant esophageal dilatation >6cm in lower esophagus
5. Disrupted mucosal integrity at the distal esophagus, eg. Ulcer, fibrotic scars etc
6. Patients with large hiatal hernias (axial length > 2 cm and Hill grade >2).
7. Patients with significant cardiorespiratory comorbidities which may limit their ability to undertake general anesthesia for the procedure, including ASA grade III or above.
8. Patients with obesity (Body Mass Index (BMI) ≥ 30).
9. Pregnant women or those planning pregnancy or breastfeeding women.
10. Uncorrectable coagulopathy defined by international normalized ratio (INR) > 1.5 or platelet count < 50000/µl.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Post-procedure rate of gastroesophageal reflux | 1 year
  Defined by updated Lyon 2.0 consensus as fulfilling one or more of the criteria:
  1. Endoscopic erosive esophagitis, LA grade B or above
  2. Long segment Barrett's esophagus
  3. Peptic esophageal stricture
  4. 24-hour pH study with acid exposure time >6% Both endoscopy and pH study to be performed with proton pump inhibitor stopped for 4 weeks

SECONDARY OUTCOMES:
Clinical success rate of procedure | 1 year
  Post-treatment Eckhardt score <=3
Adverse event of procedure | 30 day
  frequency of severe adverse events with probable or definite attribution to the procedure based on the American Society of Gastrointestinal Endoscopy (ASGE) lexicon as well as Clavien Dindo classification
Technical success rate of procedure | 1 day
  Completing all steps of the intended procedure successfully in the same session
Procedure time | 1 day
  Procedure time of the intended procedure in minutes
Erosive esophagitis on post-procedure endoscopy | 1 year
  The presence of erosive esophagitis as well as the grading on post-procedure endoscopy
Fundoplication wrap integrity on post-procedure endoscopy | 1 year
  Endoscopic appearance of fundoplication wrap on retroflexion in the stomach.
  1. Intact - wrap is completely visualised
  2. Indistinct - wrap is visualised but appears to be loosened
  3. Absent - the wrap is completely not visible
Distensibility index on EndoFLIP, premyotomy | During index procedure, before myotomy
  Distensibility index (mm2/mmHg) using EndoFLIP
Distensibility index on EndoFLIP, post myotomy | During index procedure, after myotomy
  Distensibility index (mm2/mmHg) using EndoFLIP
Distensibility index on EndoFLIP, post fundoplication | During index procedure, after fundoplication
  Distensibility index (mm2/mmHg) using EndoFLIP
Distensibility index on EndoFLIP, on follow-up | 1 year
  Distensibility index (mm2/mmHg) using EndoFLIP, at follow-up endoscopy
Maximum diameter on EndoFLIP, premyotomy | During index procedure, before myotomy
  Maximum diameter (mm) on EndoFLIP
Maximum diameter on EndoFLIP, post-myotomy | During index procedure, after myotomy
  Maximum diameter (mm) on EndoFLIP
Maximum diameter on EndoFLIP, post-fundoplication | During index procedure, after fundoplication
  Maximum diameter (mm) on EndoFLIP
Maximum diameter on EndoFLIP, on follow-up | 1 year
  Maximum diameter (mm) on EndoFLIP, at follow-up endoscopy
GERD-HRQL score | 1 month, 3 month, 6 month and 1 year
  Symptom and quality of life score relating to GERD The score ranged from 0-50 with higher score signifying more severe GERD symptom / worse quality of life
GERD-RSI score | 1 month, 3 month, 6 month and 1 year
  Symptom and quality of life score relating to GERD The score ranged from 0-45 with higher score signifying more severe GERD symptom
GERD-Q score | 1 month, 3 month, 6 month and 1 year
  Symptom and quality of life score relating to GERD The score is ranged from 0-18 with the higher score signifying more symptom of GERD
Use of proton pump inhibitor post-procedure | 1 month, 3 month, 6 month, and 1 year
  Number of participants who are on regular / as required / not on PPI

CONTACTS AND LOCATIONS:
Overall Officials: Hon Chi Yip, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (7):
- Johns Hopkins Hospital, Baltimore, Maryland, United States
- Nanfang Hospital, Southern Medical University, Guangzhou, China
- The Chinese University of Hong Kong, Hong Kong, Hong Kong
- India (4):
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Asian Institute of Gastroenterology, Hyderabad
  - Baldota Institute of Digestive Sciences, Mumbai
  - Deenanath Mangeshkar Hospital & Research Center, Pune

IPD SHARING:
Plan to Share IPD: No